CLINICAL TRIAL: NCT03362346
Title: Analysis of Physiological Signals From Neurocritical Patients in Intensive Care Units Using Wavelet Transform and Deep Learning
Brief Title: Signal Analysis for Neurocritical Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Hsin Tsai, Chief of Neurointensive Care Unit, Far Eastern Memorial Hospital
Other Study IDs: 106152-E
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Brain Injuries, Acute
Keywords: Wavelet transform; Deep learning
MeSH Terms: conditions — Brain Injuries | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurocritical patients: Patients with brain injury from trauma, ischemic stroke, hemorrhage stroke (intracerebral hemorrhage, subarachnoid hemorrhage), brain tumor with increased intracranial pressure, brain infection, hydrocephalus, among others.
  Interventions: Device: intracranial pressure monitoring

INTERVENTIONS:
Device: intracranial pressure monitoring — The patients may have either intracranial pressure (ICP) monitor insertion or external ventricular drainage that can be used as ICP monitor.
  Other Names: physiological monitoring

SUMMARY:
The project uses big data analysis techniques such as wavelet transform and deep learning to analyze physiological signals from neurocritical patients and build a model to evaluate intracranial condition and to predict neurological outcome. By identification of correlations among these parameters and their trends, we may achieve early detection of anomalies and enhance the ability in judgement of current neurological condition and prediction of prognosis. By continuous input of the past and contemporary data in the ICU, the model will be modified repeatedly and its accuracy improves as the model grows. The model can be used to recognize abnormalities earlier and provide a warning system. Clinicians taking care of neurocritical patients can adjust their treatment policy and evaluate the outcome according to such system.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or older than 20 years
* Neurocritical patients admitted to intensive care unit (ICU), including but not limited to traumatic brain injury, hemorrhagic stroke, ischemic stroke, brain infection, brain tumor and acute hydrocephalus.
* Patients who have undergone cranial surgery and had intracranial pressure monitor inserted or external ventricular drainage. The central monitor of ICU is able to collect the data continuously

Exclusion Criteria:

* Age younger than 20 years.
* Continuous monitoring of intracranial pressure is not feasible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurocritical patients admitted to intensive care unit (ICU), including but not limited to traumatic brain injury, hemorrhagic stroke, ischemic stroke, brain infection, brain tumor and acute hydrocephalus.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Neurological status | Discharge out of the intensive care unit, averaged 2 weeks
  Glasgow coma scale/Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsin Tsai, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diederik P. Kingma and Jimmy Lei Ba. Adam: A method for stochastic optimization. Conference paper at ICLR 2015.
- [Background] Michael Unser and Akram Aldroubi. (1996 Apr) A review of wavelets in biomedical applications. Proceedings of the IEEE 84(4): 626-638.
- [Background] LeCun Y, Bengio Y, Hinton G. Deep learning. Nature. 2015 May 28;521(7553):436-44. doi: 10.1038/nature14539. PMID 26017442
- [Background] Christopher Torrence and Gilbert P. Compo. (1998 Jan) A practical guide to wavelet analysis. Bulletin of the American Meteorological Society 79(1):61-78.
- [Background] Theis, Fabian & Meyer-Base, Anke. (2010). Biomedical Signal Analysis - Contemporary Methods and Applications. Biomedical Signal Analysis: Contemporary Methods and Applications.
- [Background] Min S, Lee B, Yoon S. Deep learning in bioinformatics. Brief Bioinform. 2017 Sep 1;18(5):851-869. doi: 10.1093/bib/bbw068. PMID 27473064
- [Background] Yi Mao, Wenlin Chen, Yixin Chen, Chenyang Lu, Marin Kollef, and Thomas Bailey. (2012) An integrated data mining approach to real-time clinical monitoring and deterioration warning. Proceedings of the 18th ACM SIGKDD international conference on Knowledge discovery and data mining Pages 1140-1148. doi>10.1145/2339530.2339709